CLINICAL TRIAL: NCT01630577
Title: Early Change of Central Venous Pressure With Volume Challenge as Predictor of Fluid Responsiveness in Patients With Hemodynamic Instability
Brief Title: Central Venous Pressure Change With Volume Challenge in Patients With Hemodynamic Instability
Acronym: CVPCHI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Nouira, professor, University of Monastir
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CVPChallenge
Record Dates: First submitted 2012-06-21; First posted 2012-06-28 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Acute Circulatory Failure
Keywords: acute circulatory failure; hemodynamic stability; hypovolemia
MeSH Terms: conditions — Shock; Hypovolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- responder to fluid challenge (Experimental): fluid challenge
  Interventions: Other: volume expansion using modified gelatin

INTERVENTIONS:
Other: volume expansion using modified gelatin — Volume expansion using modified gelatin was determined according to a procedure formulated by modifying guidelines produced by Weil and Henning. The maximum volume infusion during the study test was fixed at 400 ml.
  Other Names: fluid challenge

SUMMARY:
We conducted this study to assess the value of early change in central venous pressure (CVP) in predicting fluid responsiveness in mechanically ventilated patients.

DETAILED DESCRIPTION:
In patients with shock a primary goal of treatment is to restore and maintain organ perfusion, for which an adequate cardiac preload is required. Apart from the situations in which hypovolemia is evident and a favourable response to fluid administration will be seen, clinical and biological parameters often fail to predict hypovolemia. Inappropriate use of volume expansion carries out the risk of generating volume overload and pulmonary oedema. Consequently, reliable predictors of fluid responsiveness are needed especially in the early phase of cardiocirculatory deterioration. In the clinical setting, different static and dynamic indices have been shown to be useful indicators of cardiac preload. Central venous pressure (CVP) is widely used to measure right ventricular preload in patients requiring invasive hemodynamic monitoring. However, the use of the CVP is much criticized because CVP poorly predicts cardiac preload and volume status. However several decades ago, Weil and Henning proposed the fluid challenge technique, based on the 2-5 rule using CVP. There is a method for guiding volume repletion based on measurements of the patient's response to fluid load. This method has not been validated in the prediction of fluid responsiveness. We therefore conducted a prospective study that in all patients we measured CVP change and stroke volume variation (SVV) after administration of fluids. Patients were classified as fluid responders when their SVV is >10% after volume expansion and non-responders if SVV is ≤10%.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated patients
* acute circulatory failure defined by the need of vasopressive drugs (dopamine >5µg/kg/per minute or norepinephrine) with signs of tissue hypoperfusion (e.g., altered mental state, mottled skin, urine output below 0.5 ml per kilogram of body weight per hour during at least 2 h).
* admission serum lactate level more than 2.5mmol/L

Exclusion Criteria:

* severe hypoxemia defined as a ratio of arterial oxygen pressure to fraction of inspired oxygen [PaO2/FiO2] < 100 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
fluid challange responsiveness | within 20 minutes of fluid challenge
  change of Stroke volume variation (SVV) by more than 10%

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Professor, Principal Investigator — FB University Hospital Monastir Tunisia
Locations (2):
- Tunisia (2):
  - CHU Fattouma Bourguiba, Monastir, Monastir Governorate
  - Emergency Department FB University Hospital, Monastir, Monastir Governorate

IPD SHARING:
Plan to Share IPD: Undecided